CLINICAL TRIAL: NCT07231523
Title: Perioperative Efficacy and Safety of Efgartigimod Versus Intravenous Immunoglobulin for Thymoma Associated Myasthenia Gravis: a Prospective, Multicenter, Randomized Controlled Study
Brief Title: EFG vs IVIG in TAMG
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tang-Du Hospital (Other); West China Hospital (Other); Second Affiliated Hospital of Soochow University (Other); Huashan Hospital (Other); The Affiliated Brain Hospital of Nanjing Medical University (Other Government); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROMISE-TAMG
Record Dates: First submitted 2025-09-24; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Efgartigimod; Intravenous Immunoglobulin; Myasthenia Gravis Associated With Thymoma
MeSH Terms: interventions — Thymectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Efgartigimod + Thymectomy (Experimental)
  Interventions: Combination Product: Efgartigimod + Thymectomy
- Intravenous immunglobulin + Thymectomy (Active Comparator)
  Interventions: Combination Product: Intravenous immunglobulin + Thymectomy

INTERVENTIONS:
Combination Product: Efgartigimod + Thymectomy — Patients receive weight-based EFG infusions (10 mg/kg; fixed 1200 mg for ≥120 kg) administered over 1 hour once weekly for 4 total doses. If a scheduled infusion is missed, EFG may be administered within 48 hours of the planned time, followed by resumption of the original schedule to complete all 4 infusions. Thymectomy is performed on the day following the second EFG infusion with a permitted ±3-day surgical window.
  Arms: Efgartigimod + Thymectomy
Combination Product: Intravenous immunglobulin + Thymectomy — Patients receive weight-based IVIG infusions (400 mg/kg) administered daily for 5 consecutive days. Thymectomy is performed approximately 7 days after completing the final IVIG infusion, with a permitted ±3-day surgical window.
  Arms: Intravenous immunglobulin + Thymectomy

SUMMARY:
This study is a prospective, multi-center, randomized controlled study to evaluate the efficacy and safety of efgartigimod (EFG) and intravenous immunoglobulin (IVIG) in the perioperative application for acetylcholine receptor (AChR) antibody-positive thymoma patients with myasthenia gravis in order to provide reliable evidence for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged >18 years and ≤75 years, with an expected survival time >12 months;
2. Patients with generalized myasthenia gravis;
3. MG-ADL ≥6;
4. Positive for AChR antibody;
5. Diagnosed with thymoma by enhanced chest CT or MRI;
6. Patients with thymoma combined with myasthenia gravis who are diagnosed by MDT and need to undergo thymectomy;
7. Patients with American Society of Anesthesiologists (ASA) grade 1-2;
8. Able to understand the study situation and sign the Informed Consent.

Exclusion Criteria:

1. MGFA type V;
2. Patients who have undergone median sternotomy;
3. Confirmed history of congestive heart failure; poorly controlled angina pectoris with drug treatment; electrocardiogram (ECG) confirmed transmural myocardial infarction; poorly controlled hypertension; clinically significant valvular heart disease; or high-risk uncontrolled arrhythmia;
4. Patients with weight loss of more than 5kg in the past month; severe uncontrolled systemic disease, such as active infection or poorly controlled diabetes; patients with hemorrhagic diseases and bleeding tendencies; coagulation dysfunction, bleeding tendency or receiving thrombolytic or anticoagulant therapy; patients with grade II-IV bone marrow suppression;
5. Females with positive serum pregnancy test or in lactation period, and males and females of childbearing age who are unwilling to use adequate contraceptive measures during treatment;
6. History of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation);
7. Patients with peripheral nervous system disorders or significant mental disorders and a history of central nervous system disorders;
8. Patients participating in other clinical studies simultaneously;
9. Patients who cannot tolerate single-lung ventilation during surgery; severe cardiac complications, cardiovascular decompensation, patients with implanted cardiac pacemakers;
10. Patients in the acute inflammatory period due to bacterial, viral or other microbial infections; known active infections of human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV), or known HIV seropositivity;
11. Patients who have undergone thoracic surgery due to tuberculous pleurisy, mesothelioma, lung disease, or diaphragmatic disease, with ipsilateral lung atelectasis involving one lobe or more than one lobe;
12. Serum IgG level <4.5 g/L;
13. Received biological agents such as rituximab or ibritumomab tiuxetan within 6 months; underwent plasma exchange within 1 month;
14. Thrombosis, renal impairment or renal failure;
15. Allergic to human immunoglobulin or have other severe allergic history;
16. Selective IgA deficiency with anti-IgA antibodies;
17. Subjects with impaired function of major organs, abnormal blood routine, lung, liver, kidney and cardiac function, and the following laboratory test results:

Blood: white blood cells <4.0×10^9/L, absolute neutrophil count (ANC) <2.0×10^9/L, platelet count <100×10^9/L, hemoglobin <90g/L; Liver function: serum bilirubin >1.5 times the upper normal limit; ALT and AST >1.5 times the upper normal limit; Renal function: serum creatinine (SCr) >120 μmol/L, creatinine clearance rate (CCr) <60 ml/min;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative Myasthenia Gravis (QMG) reduction | From baseline to 2 weeks postoperatively
  The total QMG score ranges from 0 to 39, with higher scores indicating more severe condition.

SECONDARY OUTCOMES:
Myasthenia Gravis Activities of Daily Living (MG-ADL) reduction | From baseline to 2 weeks postoperatively
  The total MG-ADL score ranges from 0 to 24, with higher scores indicating more severe condition
Myasthenia Gravis Composite (MGC) reduction | From baseline to 2 weeks postoperatively
  The total MGC score ranges from 0 to 50, with higher scores indicating more severe condition.
QMG change (1 day preoperatively) | From baseline to 1 day preoperatively
  The change in the QMG score from baseline to 1 day preoperatively
QMG change (1 week postoperatively) | From baseline to 1 week postoperatively
  The change in the QMG score from baseline to 1 week postoperatively
QMG change (1 month postoperatively) | From baseline to 1 month postoperatively
  The change in the QMG score from baseline to 1 month postoperatively
QMG change (2 months postoperatively) | From baseline to 2 months postoperatively
  The change in the QMG score from baseline to 2 months postoperatively
MG-ADL change (1 day preoperatively) | From baseline to 1 day preoperatively
  The change in the MG-ADL score from baseline to 1 day preoperatively
MG-ADL change (1 week postoperatively) | From baseline to 1 week postoperatively
  The change in the MG-ADL score from baseline to 1 week postoperatively
MG-ADL change (1 month postoperatively) | From baseline to 1 month postoperatively
  The change in the MG-ADL score from baseline to 1 month postoperatively
MG-ADL change (2 months postoperatively) | From baseline to 2 months postoperatively
  The change in the MG-ADL score from baseline to 2 months postoperatively
MGC change (1 day preoperatively) | From baseline to 1 day preoperatively
  The change in the MGC score from baseline to 1 day preoperatively
MGC change (1 week postoperatively) | From baseline to 1 week postoperatively
  The change in the MGC score from baseline to 1 week postoperatively
MGC change (1 month postoperatively) | From baseline to 1 month postoperatively
  The change in the MGC score from baseline to 1 month postoperatively
MGC change (2 months postoperatively) | From baseline to 2 months postoperatively
  The change in the MGC score from baseline to 2 months postoperatively
IgG reduction (1 day preoperatively) | From baseline to 1 day preoperatively
  The reduction in the IgG level from baseline to 1 day preoperatively
IgG reduction (1 week postoperatively) | From baseline to 1 week postoperatively
  The reduction in the IgG level from baseline to 1 week postoperatively
IgG reduction (2 weeks postoperatively) | From baseline to 2 weeks postoperatively
  The reduction in the IgG level from baseline to 2 weeks postoperatively
IgG reduction (1 month postoperatively) | From baseline to 1 month postoperatively
  The reduction in the IgG level from baseline to 1 month postoperatively
IgG reduction (2 months postoperatively) | From baseline to 2 months postoperatively
  The reduction in the IgG level from baseline to 2 months postoperatively
AChR-Ab reduction (1 day preoperatively) | From baseline to 1 day preoperatively
  The reduction in the AChR-Ab level from baseline to 1 day preoperatively
AChR-Ab reduction (2 weeks postoperatively) | From baseline to 2 weeks postoperatively
  The reduction in the AChR-Ab level from baseline to 2 weeks postoperatively
AChR-Ab reduction (1 month postoperatively) | From baseline to 1 month postoperatively
  The reduction in the AChR-Ab level from baseline to 1 month postoperatively
Proportion of steroid dose reduction | From baseline to 2 months postoperatively
  The rate of reduction in steroid dose from baseline to 2 months postoperatively
Incidence of myasthenic crisis | Perioperative period
  The incidence of postoperative myasthenia gravis crisis, from the start of the trial to the end of the follow-up period
Incidence of total perioperative complications (≥3) | Perioperative period
  The incidence of total perioperative complications assessed by Clavien-Dindo classification
Incidence of perioperative infection-related complications | Perioperative period
  The incidence of perioperative infection-related complications assessed by Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No